CLINICAL TRIAL: NCT02824146
Title: Lung Recruitment Assessment With Lung Ultrasound In Pediatric Patient Scheduled For Abdominal Laparoscopic Surgery
Brief Title: Lung Recruitment Assessment With Lung Ultrasound In Pediatric Patient Scheduled For Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hospital Privado de Comunidad
Record Dates: First submitted 2016-06-23; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Atelectasis
Keywords: atelectasis; children; lung ultrasound; lung recruitment
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Patients received standard protective mechanical ventilation during all surgery, with tidal volumen 6 ml/kg and positive end-expiratory pressure (PEEP) level of 5 (centimeter of water) cmH2O.
- Recruitment maneuver group (Experimental): Patient received a lung recruitment maneuver after pneumoperitoneum insufflation.
  The recruitment maneuver consists in 10 breaths at 30/15 cmH2O of plateau pressure and PEEP, respectively. Then, the ventilatory settings back to protective ventilation but adding 8 cmH2O of PEEP to keep the lungs open.
  Interventions: Other: Lung recruitment maneuver

INTERVENTIONS:
Other: Lung recruitment maneuver — The lung recruitment maneuver consists in a brief and controlled increment in airways pressure (15 cmH2O of PEEP + 15 cmH2O of driving pressure) for 10 breaths.
  Arms: Recruitment maneuver group

SUMMARY:
Anesthesia-induced atelectasis is a well-known entity observed in approximately 68-100% of pediatric patients undergoing general anesthesia. The collapse of dependent lung zones starts with anesthesia induction but can persist for hours or even days after surgery. Such anesthesia-related atelectasis has a number of negative clinical consequences such as the impairment of arterial blood oxygenation and lung mechanics as well as the predisposition for ventilator-associated lung injury. The adjustment of ventilator settings for preventing the occurrence of atelectasis and for reducing pulmonary complications remains controversial.

Lung sonography (LUS) plays an important role in diagnosing pulmonary diseases in children, including atelectasis of different origins. LUS has demonstrated its high sensitivity and specificity for diagnosing anesthesia-induced atelectasis in children.

DETAILED DESCRIPTION:
Compare lung aeration between two different mechanical ventilation strategies (protective mechanical ventilation and recruitment maneuvers) in pediatric patients scheduled for abdominal laparoscopic surgery using ultrasound imaging and a four-point-aeration score to assess the lung aeration.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by parents.
* Patients aged 6 months to 7 years old
* Scheduled for abdominal laparoscopic surgery
* American Society of Anesthesiologists classification: physical status I-II

Exclusion Criteria:

* Acute airway infection
* Cardiovascular and or pulmonary disease
* Previous thoracic procedure

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Compare lung aeration between protective mechanical ventilation and recruitment maneuvers in pediatric patients scheduled for abdominal laparoscopic surgery using ultrasound imaging and a four point aeration score to assess the lung aeration | intraoperative
  Compare lung aeration between protective mechanical ventilation and recruitment maneuvers in pediatric patients scheduled for abdominal laparoscopic surgery using ultrasound imaging and a four point aeration score (0: normal lung aeration, 1: moderate loss of lung aeration, 2: severe loss of lung aeration, 3: complete loss of lung aeration and lung consolidation).

SECONDARY OUTCOMES:
Lung aeration score pre/post the recruitment maneuver during laparoscopic surgery | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Maria Acosta, MD, Principal Investigator — Hospital Privado de Comunidad

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376
- [Background] Serafini G, Cornara G, Cavalloro F, Mori A, Dore R, Marraro G, Braschi A. Pulmonary atelectasis during paediatric anaesthesia: CT scan evaluation and effect of positive endexpiratory pressure (PEEP). Paediatr Anaesth. 1999;9(3):225-8. doi: 10.1046/j.1460-9592.1999.00340.x. PMID 10320601
- [Background] Tusman G, Bohm SH, Vazquez de Anda GF, do Campo JL, Lachmann B. 'Alveolar recruitment strategy' improves arterial oxygenation during general anaesthesia. Br J Anaesth. 1999 Jan;82(1):8-13. doi: 10.1093/bja/82.1.8. PMID 10325828
- [Derived] Acosta CM, Sara T, Carpinella M, Volpicelli G, Ricci L, Poliotto S, Abrego D, Gonorazky S, Bohm SH, Tusman G. Lung recruitment prevents collapse during laparoscopy in children: A randomised controlled trial. Eur J Anaesthesiol. 2018 Aug;35(8):573-580. doi: 10.1097/EJA.0000000000000761. PMID 29278555